CLINICAL TRIAL: NCT01395563
Title: Strength Training on Pancreatic Cancer
Acronym: STOPC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: Heidelberg University (Other); Technical University of Munich (Other)
Responsible Party: Krakowski-Roosen, Dr., German Cancer Research Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GermanCRC
Record Dates: First submitted 2009-12-04; First posted 2011-07-15 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Pancreatic Neoplasms; Cachexia; Myopathy
MeSH Terms: conditions — Pancreatic Neoplasms; Cachexia; Muscular Diseases | interventions — Resistance Training; dermcidin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): pancreatic cancer patients
  Interventions: Behavioral: strength training
- 2 (Experimental): pancreatic cancer patients
  Interventions: Behavioral: strength training

INTERVENTIONS:
Behavioral: strength training — strength training, high intensity, twice up to 3 times per week
  Other Names: progressive resistance training; sports; muscle hypertrophia; cachexia

SUMMARY:
The purpose of this study is to determine whether prednisone, methotrexate, and cyclophosphamide are effective in the treatment of rapidly progressive hearing loss in both ears due to autoimmune inner ear disease (AIED).

DETAILED DESCRIPTION:
Sudden out-of-hospital cardiac arrest (OOH-CA) remains a significant cause of death, in spite of recent declines in overall mortality from cardiovascular disease. Existing methods of emergency resuscitation are inadequate due to time delays inherent in the transport of a trained responder with defibrillation capabilities to the side of the OOH-CA victim. Existing Emergency Medical Services (EMS) systems typically combine paramedic Emergency Medical Technician (EMT) services with some level of community involvement, such as bystander cardiopulmonary resuscitation (CPR) training. Some communities include automated external defibrillators (AEDs) at isolated sites or in mobile police or fire vehicles. A comprehensive, integrated community approach to treatment with AEDs would have community units served by these volunteer non-medical responders who can quickly identify and treat a patient with OOH-CA. Such an approach is termed Public Access Defibrillation (PAD).

ELIGIBILITY:
Inclusion Criteria:

* patients with pancreatic carcinomas after surgery (resection or exploration)
* given consent

Exclusion Criteria:

* acute infection
* pain
* no mobility or ability for walking or standing
* severe neurological disorders (apoplex, morbus Parkinson, paresis of the lower extremeties)
* severe cardiac or cardiovascular diseases (z.B. heart insufficiency NYHA III, myocardial infarction <3 months)
* rhytmical disorders, that contraindicate ergospirometric examinations
* cardiac therapy with digitalis pharmacy
* unclear syncopes
* severe pulmonal insufficiency
* renal insufficiency (GFR < 30% at Krea >3 mg/dl)
* synchronous participation in an other clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
muscle mass and strength | after 8 weeks of intervention

SECONDARY OUTCOMES:
quality of life | after 8 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jens Werner, Prof. Dr. med., Principal Investigator — Heidelberg University; Holger Krakowski-Roosen, Dr., Principal Investigator — German CRC; Marc Martignoni, PD Dr. med., Principal Investigator — Technical University of Munich
Locations (3):
- Germany (3):
  - European Pancreas Center, Heidelberg
  - German Cancer Research Center, Heidelberg
  - Technische Universität München, Munich